CLINICAL TRIAL: NCT00596336
Title: A Randomized Phase II Trial to Determine Whether the Application of Imiquimod Cream to the Vaccination Site Can Improve the Immune Responsiveness to Influenza Vaccination in Patients With Untreated Chronic Lymphocytic Leukemia
Brief Title: Study of Immune Responses to Influenza Vaccination With or Without Imiquimod Application in Untreated CLL Patients
Acronym: CLLIFVAC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: The Royal Bournemouth Hospital (Other)
Collaborators: CLL Topics, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: Eudract number: 2006-004902-16; LREC number: 06/Q2201/143
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A CLL patients (Active Comparator): Vaccination with current trispecific influenza vaccine Day 1
  Interventions: Drug: influenza vaccine
- Group B CLL patients (Experimental): Vaccination with current trispecific influenza vaccine Day 1, together with the application of Imiquimod cream to the vaccination site on day 2 to 6.
  Interventions: Drug: Imiquimod cream; Drug: influenza vaccine
- Group C volunteers (Active Comparator): Vaccination with current trispecific influenza vaccine Day 1
  Interventions: Drug: influenza vaccine

INTERVENTIONS:
Drug: Imiquimod cream — Imiquimod (aldara) 0.5 % cream to site of vaccination on day 2 to 6
  Other Names: Aldara cream
  Arms: Group B CLL patients
Drug: influenza vaccine — trispecific influenza vaccine 0.5 ml subcutaneously
  Other Names: influvac sub-unit

SUMMARY:
The purpose of the study is to determine whether it is possible to improve the immune response rate to 'flu vaccination in patients with chronic lymphocytic leukaemia (CLL).

Annual flu vaccination is recommended for all patients with CLL because they are known to be susceptible to infections and particularly to chest infections that may occur as a complication of influenza. Protection against 'flu depends on patients having a high level of antibodies against the 'flu virus. Vaccination works by stimulating the immune system and thus boosting the levels of these protective antibodies.

CLL patients have weakened immune systems due to the leukaemia itself but also following chemotherapy. The exact cause of these immune defects is not known. However, CLL patients typically have low antibody levels and their immune cells may not work normally.

Unfortunately, studies have shown that patients with CLL are not very good at making antibodies to 'flu vaccination and as a result protection against flu is not very reliable. Recent studies have shown that only 15-20 % of CLL patients will achieve a protective antibody level.

Recently a new type of medical cream has been introduced to treat certain skin conditions. Its name is Imiquimod and it is licensed to treat viral warts in the genital area and a type of skin cancer called basal cell carcinoma. It works by increasing the immune response in the skin. Animal studies have shown that as well as increasing immunity against viruses and cancers, it increases responses to vaccination when applied at the site of vaccination.

In this study we propose to test whether this new medicine can improve the response to the 'flu jab.

DETAILED DESCRIPTION:
Trial Summary

68 patients with stage A CLL who have not been treated, and 34 healthy age and sex matched volunteers who fulfil the entry requirements will be identified and invited to take part in this study.

Blood samples will be taken for baseline studies [FBC, U&E, LFT, Immunoglobulins (Igs), haemagglutinin titres] (20 mls) and T cells studies (50 mls to be frozen).If CLL prognostic factors have not already been determined a further 20ml will be taken for these.

Patients will be randomized to either:

Group A Vaccination with current trispecific influenza vaccine Day 1

or

Group B Vaccination with current trispecific influenza vaccine Day 1, together with the application of Imiquimod cream to the vaccination site on day 2 to 6.

Blood samples will be taken on day 0 for haemagglutinin studies (20 ml) and T cells (50ml to be frozen), then on day 7, 14 for T-cell studies (50 ml) and day 28 for haemagglutinin studies (20 ml). During the 28 days that subjects participate in the trial approximately 190 ml will be taken in total.

Antibody and T-cell responses to influenza virus will be assessed and compared between the two patient arms of the study and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Untreated stage A CLL patients
* Healthy volunteers

Exclusion Criteria:

* Patients with other malignancies
* Patients receiving corticosteroids or other immunosuppressive drugs
* Patients who have received vaccination against influenza in the past 6 months
* Patients who have had an allergic reaction to a flu shot in the past, or have an allergy to eggs or who previously developed Guillain-Barré syndrome within 6 weeks of getting a flu shot
* Patients failing to give informed consent.
* Patients using homeopathic remedies such as echniaea cream.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-10; Primary Completion 2011-12 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Immune responses to influenza vaccine in CLL cohorts and healthy age matched controls | Dec 2009

SECONDARY OUTCOMES:
Investigate immune responses and correlate with CLL prognostic markers | Dec 2009

CONTACTS AND LOCATIONS:
Overall Officials: Helen McCarthy, MBBS PhD, Principal Investigator — Royal Bournemouth Hospital
Locations (1):
- Royal Bournemouth hospital, Bournemouth, Dorset, United Kingdom